CLINICAL TRIAL: NCT00708435
Title: An Open-label, Randomized, Multicenter Phase IIIb Study to Assess the Efficacy, Safety and Tolerance of BERIPLEX® P/N Compared With Plasma for Rapid Reversal of Coagulopathy Induced by Coumarin Derivatives in Subjects With Acute Major Bleeding
Brief Title: Efficacy and Safety Study of BERIPLEX® P/N (Kcentra) Compared With Plasma in Patients With Acute Major Bleeding Caused by Anticoagulant Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE1116_3002; 1462 (Other: CSL Behring); 2007-007861-19 (EudraCT Number)
Record Dates: First submitted 2008-07-01; First posted 2008-07-02 (Estimated); Results first posted 2013-08-13 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2013-09

CONDITIONS: Blood Coagulation Disorders; Acute Major Bleeding
Keywords: Anticoagulant reversal; Prothrombin; Complex; Concentrate; Coagulopathy; induced by; coumarin; derivatives; Kcentra
MeSH Terms: conditions — Blood Coagulation Disorders; Hemostatic Disorders

ARMS (2):
- Beriplex® P/N (Experimental)
  Interventions: Biological: Beriplex® P/N (Kcentra)
- Fresh frozen plasma (Active Comparator)
  Interventions: Biological: Fresh frozen plasma

INTERVENTIONS:
Biological: Beriplex® P/N (Kcentra) — Intravenous infusion, dosage depending on baseline INR, amount of coagulation factor IX and body weight
  Other Names: Kcentra
  Arms: Beriplex® P/N
Biological: Fresh frozen plasma — Intravenous Infusion, dosage depending on baseline INR and body weight
  Arms: Fresh frozen plasma

SUMMARY:
The purpose of this study is to evaluate efficacy, safety and tolerance of BERIPLEX® P/N (Kcentra) compared with plasma in regard to rapid reversal of coagulopathy induced by coumarin derivatives in subjects who require immediate correction of INR (International Normalized Ratio)and to stop an acute major bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 years
* Subjects who have received oral vitamin K-antagonist therapy
* Subjects who have acute major bleeding, defined as one of the following: life-threatening or potentially life-threatening, acute bleeding associated with a fall in hemoglobin (Hb) level ≥ 2g/dL, bleeding requiring blood product transfusion
* INR ≥ 2 within 3 hours before start of study treatment
* Informed consent has been obtained

Exclusion Criteria:

* Expected survival of less than 3 days, or expected surgery in less than 1 day
* Acute trauma for which reversal of vitamin K antagonists alone would not be expected to control the acute bleeding event
* Use of unfractionated or low molecular weight heparin use from 24 hours prior to enrollment or expected need within 24 hours after start of infusion
* For patients with ICH: Glasgow coma score (GCS) < 7; intracerebral hematoma volume > 30cc as assessed by ABC/21; for subdural hematomas: maximum thickness ≥ 10 mm, midline shift ≥ 5 mm; for subarachnoid hemorrhage: any evidence of hydrocephalus; infratentorial ICH location; epidural hematomas; intraventricular extension of hemorrhage; modified Rankin score (mRS) of >3 prior to ICH
* History of thrombotic event, myocardial infarction, disseminated intravascular coagulation, cerebral vascular accident, transient ischemic attack, unstable angina pectoris, or severe peripheral vascular disease within 3 months of enrollment
* Known history of antiphospholipid antibody syndrome or lupus anticoagulant antibodies
* Suspected or confirmed sepsis at time of enrollment
* Administration of whole blood, plasma, plasma fractions or platelets within 2 weeks prior to inclusion into the study
* Large blood vessel rupture (e.g. in advanced cancer patient)
* Pre-existing progressive fatal disease with a life expectancy of less than 2 months
* Known inhibitors to coagulation factors II, VII, IX, or X; or hereditary protein C or protein S deficiency; or heparin-induced, type II thrombocytopenia
* Treatment with any other investigational medicinal product within 30 days prior to inclusion into the study
* Presence or history of hypersensitivity to components of the study medication
* Pregnant or breast-feeding women
* Prior inclusion in this study or any other CSL Behring-sponsored Beriplex study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring
Locations (65):
- United States (37):
  - Study Site, Birmingham, Alabama
  - Study Site, Los Angeles, California
  - Study Site, San Franciso, California
  - Study Site, Newark, Delaware
  - Study Site, Orlando, Florida
  - Study Site, Tampa, Florida
  - Study Site, Chicago, Illinois
  - Study Site, Oak Park, Illinois
  - Study Site, Hazard, Kentucky
  - Study Site, Baltimore, Maryland
  - Study Site, Boston, Massachusetts
  - Study Site, Worchester, Massachusetts
  - Study Site, Ann Arbor, Michigan
  - Study Site, Royal Oak, Michigan
  - Study Site, Duluth, Minnesota
  - Study Site, Minneapolis, Minnesota
  - Study Site, Jackson, Mississippi
  - Study Site, St Louis, Missouri
  - Study Site, Albuquerque, New Mexico
  - Study Site, Albany, New York
  - Study Site, Johnson City, New York
  - Study Site, New York, New York
  - Study Site, Rochester, New York
  - Study Site, Staten Island, New York
  - Study Site, Durham, North Carolina
  - Study Site, Allentown, Pennsylvania
  - Study Site, Hershey, Pennsylvania
  - Study Site, Philadelphia, Pennsylvania
  - Study Site, West Reading, Pennsylvania
  - Study Site, Austin, Texas
  - Study Site, El Paso, Texas
  - Study Site 2, Houston, Texas
  - Study Site, Houston, Texas
  - Study Site, Temple, Texas
  - Study Site, Salt Lake City, Utah
  - Study Site, Charlottesville, Virginia
  - Study Site, Richmond, Virginia
- Belarus (2):
  - Study Site 1, Minsk
  - Study Site 2, Minsk
- Bulgaria (7):
  - Study Site, Pleven
  - Study Site, Plovdiv
  - Study Site, Rousse
  - Study Site 1, Sofia
  - Study Site 2, Sofia
  - Study Site 3, Sofia
  - Study Site 4, Sofia
- Romania (6):
  - Study Site, Brasov
  - Study Site 1, Bucharest
  - Study Site 2, Bucharest
  - Study Site 3, Bucharest
  - Study Site, Cluj-Napoca
  - Study Site, Timișoara
- Russia (11):
  - Study Site, Arkhangelsk
  - Study Site 1, Barnaul
  - Study Site 2, Barnaul
  - Study Site, Kazan'
  - Study Site, Kemerovo
  - Study Site 1, Moscow
  - Study Site 2, Moscow
  - Study Site 1, Nizhny Novgorod
  - Study Site 2, Nizhny Novgorod
  - Study Site 1, Saint Petersburg
  - Study Site 2, Saint Petersburg
- Ukraine (2):
  - Study Site, Kharkiv
  - Study Site, Vinnytsa

REFERENCES:
- [Result] Sarode R, Milling TJ Jr, Refaai MA, Mangione A, Schneider A, Durn BL, Goldstein JN. Efficacy and safety of a 4-factor prothrombin complex concentrate in patients on vitamin K antagonists presenting with major bleeding: a randomized, plasma-controlled, phase IIIb study. Circulation. 2013 Sep 10;128(11):1234-43. doi: 10.1161/CIRCULATIONAHA.113.002283. Epub 2013 Aug 9. PMID 23935011

RESULTS

PARTICIPANT FLOW:
Groups:
- Beriplex® P/N: Beriplex® P/N : Single intravenous infusion as required to treat acute major bleeding; dosage 25, 35 or 50 units/kg depending on baseline INR, amount of coagulation factor IX and body weight.
- Fresh Frozen Plasma: Fresh frozen plasma : Single intravenous infusion as required to treat acute major bleeding; dosage 10, 12, or 15 mL/kg depending on baseline INR and body weight.
Period: Overall Study
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Started | 107 | 109
Completed | 82 (These data are 'on-study' results collected up to the subject's Day 45 visit.) | 92 (These data are 'on-study' results collected up to the subject's Day 45 visit.)
Not Completed | 25 | 17
Not completed — Death / Serious Adverse Event | 10 | 5
Not completed — Lost to Follow-up | 9 | 4
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Intervention by primary care physician | 1 | 0
Not completed — Refused hospitalization | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intention-to-treat population comprised all subjects who were (1) eligible for the study and had (2) signed informed consent and were randomized to 1 of the 2 treatment groups regardless of whether the subjects received study product. In the ITT population, subjects were analyzed "as randomized".
Groups:
- Beriplex® P/N: Beriplex® P/N : Intravenous infusion, dosage depending on baseline INR, amount of coagulation factor IX and body weight
- Fresh Frozen Plasma: Fresh frozen plasma : Intravenous Infusion, dosage depending on baseline INR and body weight
- Total: Total of all reporting groups
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma | Total
Number analyzed (Participants) | 107 | 109 | 216
Age, Customized [Number; unit: Participants]
  < 65 years | 36 | 32 | 68
  ≥ 65 to < 75 years | 28 | 29 | 57
  ≥ 75 years | 43 | 48 | 91
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 55 | 107
  Male | 55 | 54 | 109

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hemostatic Efficacy of Stopping an Ongoing Major Bleed
Description: Hemostatic efficacy was determined by a blinded independent board as excellent, good, or poor/none, based on prespecified definitions. Assessments of visible or non-visible musculoskeletal bleeding were made at 1 and 4 hours after the end of infusion. Hemostatic efficacy was the binary endpoint of effective or non-effective hemostasis, where 'effective' was a hemostatic efficacy rating of "excellent" or "good," and 'non-effective' was a hemostatic efficacy rating of "poor/none".
Time Frame: At 1 and 4 hours after the end of infusion
Population: The Intention-to-Treat Efficacy (ITT-E) population included all randomized participants who had received any study product, presented with acute major bleeding, and had an international normalized ratio (INR) > 1.3 prior to the infusion. Participants in the ITT-E population were analyzed 'as randomized'.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Beriplex® P/N: Beriplex® P/N: Intravenous infusion, dosage depending on baseline INR, amount of coagulation factor IX and body weight
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 98 | 104
percentage of participants | 72.4 [63.6 to 81.3] | 65.4 [56.2 to 74.5]
Statistical Analysis 1: Comparison: Beriplex® P/N vs Fresh Frozen Plasma; The analysis of hemostatic efficacy was via calculation of the 95% confidence interval (CI) for the difference (Beriplex minus plasma) in the percentage of participants with effective hemostasis; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was -(minus)10%. If the lower limit of the 2-sided 95% CI was >-10%, then the null-hypothesis was rejected and it was concluded that Beriplex was non-inferior to plasma. The sample size estimation assumed that hemostatic efficacy would be rated 'effective' in 85% of participants in the plasma group and 90% of participants in the Beriplex group. The power to show non-inferiority with these assumptions was greater than 80% for two treatment groups of 83 participants; 95% confidence interval — Both primary endpoints had to be non-inferior for Beriplex to be non-inferior. No P-value is entered as non-inferiority was assessed via the 95% CI calculation for the difference (Beriplex minus plasma) in the % of subjects with effective hemostasis; Farrington and Manning's method was used to estimate the 95% CI for the difference in the percentage of participants with hemostasis; Difference in effective hemostasis (%) = 7.1, 95% CI 2-sided [-5.8 to 19.9] — Both primary endpoints had to be non-inferior for Beriplex to be non-inferior. There is no P-value as non-inferiority was assessed via the 95% CI calculation for the difference (Beriplex minus plasma) in the % of subjects with effective hemostasis

2. Primary Outcome: Percentage of Participants Who Had a Rapid Decrease of the International Normalized Ratio (INR)
Description: A rapid decrease of the international normalized ratio (INR) was defined as an INR ≤ 1.3 at 30 minutes after the end of the infusion. The INR is a standard way to describe the time it takes for blood to clot; an INR range of 0.8 to 1.2 is considered normal for a healthy person who is not using oral anticoagulant therapy.
Time Frame: 30 minutes after end of infusion
Population: The ITT-E population included all randomized participants who had received any study product, presented with acute major bleeding, and had an INR > 1.3 prior to the infusion. Participants in the ITT-E population were analyzed 'as randomized'.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 98 | 104
percentage of participants | 62.2 [52.6 to 71.8] | 9.6 [3.9 to 15.3]
Statistical Analysis 1: Comparison: Beriplex® P/N vs Fresh Frozen Plasma; The analysis of the percentage of participants who had a rapid decrease of the INR was via calculation of the 95% confidence interval (CI) for the difference (Beriplex minus plasma) in the percentage of participants with a rapid decrease of the INR; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; 95% confidence interval — Both primary endpoints had to be non-inferior for Beriplex to be non-inferior. No P-value is entered as non-inferiority was assessed via the 95% CI for the difference (Beriplex minus plasma) in the % of subjects with a rapid decrease of the INR; Farrington and Manning's method was used to estimate the 95% CI for the difference in the percentage of participants with a rapid decrease of the INR; Difference in the decrease of INR (%) = 52.6, 95% CI 2-sided [39.4 to 65.9] — Both primary endpoints had to be non-inferior for Beriplex to be non-inferior. There is no P-value as non-inferiority was assessed via the 95% CI for the difference (Beriplex minus plasma) in the % of subjects with a rapid decrease of the INR

3. Secondary Outcome: Percentage of Participants Who Had Hemostatic Efficacy for Visible or Non-visible Musculoskeletal Bleeding
Description: Hemostatic efficacy was determined by a blinded independent board as excellent, good, or poor/none, based on prespecified definitions. Assessments of visible or non-visible musculoskeletal bleeding were made at 3 and 6 hours after the start of infusion. Hemostatic efficacy was the binary endpoint of effective or non-effective hemostasis, where 'effective' was a hemostatic efficacy rating of "excellent" or "good," and 'non-effective' was a hemostatic efficacy rating of "poor/none".
Time Frame: At 3 and 6 hours after the start of infusion
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 98 | 104
percentage of participants | 73.5 [64.7 to 82.2] | 67.3 [58.3 to 76.3]

4. Secondary Outcome: Incremental in Vivo Recovery (IVR) (Response) of Factors II, VII, IX, and X, Protein C, and Protein S for Beriplex
Description: The incremental IVR [(IU/dL)/(IU/kg)] was calculated as follows: (IU/dL activity rise in plasma)/(IU/kg body weight infused) = [maximum increase in component plasma level within 3 hours compared to pre-infusion (IU/dL)]/{[exact dose of component in drug administered (IU)]/[body weight (kg)]}.
Time Frame: Before infusion and up to 3 h after the start of infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg body weight)
Arm/Group | Beriplex® P/N
Number analyzed (Participants) | 97
(IU/dL)/(IU/kg body weight)
  Factor II | 2.00 (0.879)
  Factor VII | 2.15 (2.958)
  Factor IX | 1.29 (0.711)
  Factor X | 1.96 (0.871)
  Protein C | 2.04 (0.958)
  Protein S | 2.17 (1.661)

5. Secondary Outcome: Plasma Levels of Factors II, VII, IX, and X, Protein C, and Protein S
Description: Plasma levels are presented as the percentage of normal at pre-infusion and 30 min and 24 h after the start of infusion. The plasma level assay results are reported as a potency relative to a standard, where 100% is considered to be normal.
Time Frame: From preinfusion until 24 h after the start of infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of normal
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 98 | 104
percentage of normal
  Factor II, pre-infusion (n = 98; 103) | 20.1 (14.56) | 22.3 (22.39)
  Factor II, 0.5 h after infusion start (n = 88; 90) | 87.5 (44.48) | 31.9 (22.55)
  Factor II, 24 h after infusion start (n = 92; 99) | 77.1 (22.06) | 58.1 (19.55)
  Factor VII, pre-infusion (n = 98; 103) | 25.9 (35.01) | 23.5 (23.45)
  Factor VII, 0.5h after infusion start (n = 88; 90) | 60.5 (45.23) | 34.6 (26.18)
  Factor VII, 24 h after infusion start (n = 92; 99) | 114.8 (165.28) | 101.3 (79.01)
  Factor IX, pre-infusion (n = 98; 103) | 36.1 (22.56) | 39.0 (27.56)
  Factor IX, 0.5 h after infusion start (n = 88; 90) | 76.8 (35.47) | 47.7 (26.78)
  Factor IX, 24 h after infusion start (n = 92; 99) | 88.5 (35.65) | 93.0 (29.95)
  Factor X, pre-infusion (n = 98; 102) | 13.0 (11.25) | 14.7 (18.83)
  Factor X, 0.5 h after infusion start (n = 88; 90) | 99.8 (56.07) | 23.9 (20.40)
  Factor X, 24 h after infusion start (n = 92; 99) | 83.7 (27.05) | 58.2 (21.78)
  Protein C, pre-infusion (n = 98; 103) | 39.3 (17.15) | 41.1 (18.84)
  Protein C, 0.5 h after infusion start (n = 88; 90) | 110.3 (47.37) | 50.9 (24.78)
  Protein C, 24h after infusion start (n = 92; 98) | 90.3 (27.19) | 82.8 (24.34)
  Protein S, pre-infusion (n = 97; 102) | 27.8 (11.34) | 29.6 (12.97)
  Protein S, 0.5 h after infusion start (n = 88; 89) | 59.4 (28.56) | 38.6 (20.45)
  Protein S, 24 h after infusion start (n = 91; 97) | 47.8 (16.54) | 45.4 (16.00)

6. Secondary Outcome: Percentage of Participants With INR Correction at Various Times After the Start of Infusion
Description: The time taken from the start of infusion to INR correction (defined as an INR ≤ 1.3) was recorded. The percentage of participants with INR correction was calculated at 0.5, 1, 3, 6, 12, and 24 h after the start of infusion.
Time Frame: From the start of infusion until INR correction; calculated at 0.5, 1, 3, 6, 12, and 24 h after the start of infusion.
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 98 | 104
percentage of participants
  0.5 h | 4 | 0
  1 h | 69 | 0
  3 h | 71 | 9
  6 h | 78 | 16
  12 h | 80 | 36
  24 h | 88 | 58

7. Secondary Outcome: Percentage of Participants With INR Correction at Various Times After Randomization
Description: The time taken from randomization to INR correction (defined as an INR ≤ 1.3) was recorded. The percentage of participants with INR correction was calculated at 2.5, 3, 5, 8, 14, and 26 h after randomization.
Time Frame: From randomization until INR correction; calculated at 2.5, 3, 5, 8, 14, and 26 h after randomization.
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 98 | 104
percentage of participants
  2.5 h | 59 | 2
  3 h | 67 | 2
  5 h | 76 | 10
  8 h | 79 | 22
  14 h | 84 | 38
  26 h | 90 | 70

8. Secondary Outcome: Transfusion of Red Blood Cells
Description: Red blood cells were packed red blood cells (PRBCs).
Time Frame: From the start of infusion until 24 h after the start of infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units of PRBCs
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 98 | 104
Units of PRBCs | 1.4 (1.77) | 1.2 (1.57)

9. Secondary Outcome: Use of Other Blood Products and Hemostatic Agents
Description: Other blood products and hemostatic agents containing coagulation factors (such as whole blood, plasma, albumin, platelets) not including PRBCs.
Time Frame: From the start of infusion until 24 h after the start of infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units of blood products
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 98 | 104
Units of blood products | 0.3 (1.36) | 0.3 (0.87)

10. Secondary Outcome: 45-Day All-cause Mortality
Time Frame: Until Day 45
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 98 | 104
participants | 9 | 5

11. Secondary Outcome: Overall Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs. Treatment-related AEs were defined as events whose relationship to study treatment was definitely related, probably related, or possibly related in the opinion of the investigator. AEs with missing relationship were considered related to treatment. Serious TEAEs were treatment-emergent SAEs. Deaths reported up to and including Day 45; one additional Beriplex death occurred after Day 45.
Time Frame: From the start of infusion up to the allowed time window of the Day 10 visit for non-serious AEs and from the start of infusion up to the allowed time window of the Day 45 visit for SAEs.
Population: The ITT-S population included all participants who were randomized and who had received any portion of study product. Participants in the ITT-S population were analyzed 'as treated'.
Measure: Number; unit: participants
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Number analyzed (Participants) | 103 | 109
participants
  Any TEAE | 66 | 71
  At least possibly treatment-related TEAE | 10 | 23
  Serious TEAE | 32 | 26
  Death | 10 | 5

ADVERSE EVENTS:
Time Frame: From the start of infusion up to the allowed time window of the Day 45 visit for SAEs, and from the start of infusion up to the allowed time window of the Day 10 visit for non-serious AEs.
Description: The AEs presented were treatment-emergent AEs (TEAEs). The ITT-S population included all subjects who were randomized and who had received any portion of study product. Participants in the ITT-S population were analyzed 'as treated'. "General disorders" were collected under the MedDRA SOC General disorders and administration site conditions.
Arm/Group | Beriplex® P/N | Fresh Frozen Plasma
Serious Adverse Events (participants affected / at risk) | 32/103 | 26/109
Other Adverse Events (participants affected / at risk) | 46/103 | 40/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Beriplex® P/N (N=103) | Fresh Frozen Plasma (N=109)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Device dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 4 (5)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Beriplex® P/N (N=103) | Fresh Frozen Plasma (N=109)
Oedema peripheral (General disorders) | 6 (6) | 7 (7)
Pyrexia (General disorders) | 4 (4) | 4 (4)
Chest pain (General disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 10 (10) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Tachycardia (Cardiac disorders) | 4 (4) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
International normalised ratio increased (Investigations) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 3 (3)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2)
Agitation (Psychiatric disorders) | 3 (3) | 1 (1)
Mental status change (Psychiatric disorders) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Hypotension (Vascular disorders) | 5 (5) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.